CLINICAL TRIAL: NCT06768125
Title: Hypofractionated Radiotherapy for Squamous Cell Carcinoma of the Head and Neck in Elderly Patients: A Prospective Phase II Clinical Study
Brief Title: Hypofractionated Radiotherapy for HNSCC in Elderly Patients
Acronym: HNSCC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4265
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma; ELDERLY PEOPLE; Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypofractionated radiation (Experimental): The hypofractionated radiotherapy regimen specified in this study is as follows:
  Radiotherapy: The positioning is referenced from the guidelines of the Radiation Oncology Department of the Chinese Academy of Medical Sciences Cancer Hospital. The specific contouring and target area definitions are provided in the main text. The recommended radiation doses and fractionation methods are:
  95% PGTVp: 33 Gy in 3.3 Gy per session for 10 sessions, and 95% PTV1: 25 Gy in 1.5 Gy per session for 10 sessions, with an interval of 1-2 weeks, for a total of 2 cycles.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — 95% PGTVp: 33 Gy in 3.3 Gy per session for 10 sessions, and 95% PTV1: 25 Gy in 1.5 Gy per session for 10 sessions, with an interval of 1-2 weeks, for a total of 2 cycles.

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is a common malignant tumor, with 25% of HNSCC patients diagnosed at over 70 years of age. As the population ages, it is expected that by 2030, this proportion will exceed 60%. Elderly patients are gradually becoming the main population among head and neck cancer patients. Older patients often have a lower desire to seek medical treatment, leading to a higher number of late-stage diagnoses. Additionally, with declining physical function and multiple comorbidities, frequent hospital visits can be inconvenient, making them often unsuitable for aggressive surgery or comprehensive treatment.

In clinical practice, the commonly used conventional fractionated radiotherapy (66-70 Gy in 1.8-2.2 Gy per session over 30-33 sessions, completed in 6-7 weeks) is a time-consuming and intensive treatment method, often resulting in significant and prolonged acute and late toxicities. Hypofractionated radiotherapy (HFRT) significantly reduces the number of treatment sessions and shortens the treatment duration compared to conventional fractionation. Additionally, delivering higher doses can quickly and effectively reduce tumor burden by increasing the lethality to tumor cells.

Currently, there are few reports on HFRT for head and neck cancer patients abroad, and no reports on this treatment regimen for elderly HNSCC patients in China. In preliminary studies, our research group utilized a segmented hypofractionated regimen (66 Gy in 3.3 Gy per session for 20 sessions, treated for 2 weeks, followed by 1 week of rest, and then treated for another 2 weeks) to treat 12 HNSCC patients aged 77 to 97 years. The recent effective rate was 100%, with good treatment tolerance and no severe toxic reactions observed.

DETAILED DESCRIPTION:
This study aims to conduct a prospective study to evaluate the efficacy and safety of segmented hypofractionated radiotherapy in elderly patients with head and neck squamous cell carcinoma and to explore a radiotherapy fractionation scheme suitable for elderly HNSCC patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years;
2. Patients with histologically or cytologically confirmed stage II-IVA head and neck squamous cell carcinoma (AJCC 8th edition), including oral cavity, oropharynx, hypopharynx, larynx, and cervical metastatic squamous carcinoma of unknown primary;
3. At least one measurable lesion;
4. No prior systemic antitumor treatment or locoregional therapy for head and neck squamous cell carcinoma;
5. ECOG performance status of 1-3;
6. Expected survival time of ≥ 3 months;
7. Patients assessed by the physician as unsuitable for surgical treatment and not candidates for radical radiotherapy;
8. Functional status of vital organs compatible with daily basic activities (excluding any blood components or cell growth factors within 14 days): adequate bone marrow reserve function: white blood cells (WBC) ≥ 2.0 × 10^9/L, neutrophil count (NEUT) ≥ 1.0 × 10^9/L, platelet count (PLT) ≥ 80 × 10^9/L, hemoglobin (Hb) ≥ 90 g/L;
9. Able and willing to comply with the study and follow-up procedures;
10. The subject voluntarily agrees to participate in this clinical study and signs the informed consent form, demonstrating good compliance and ability to cooperate with follow-up.

Exclusion Criteria:

1. Previously undergone radiotherapy for head and neck cancer;
2. Squamous cell carcinoma of other primary sites in the head and neck, such as paranasal sinuses, nasopharynx, glottic laryngeal cancer, skin, or salivary gland tissues;
3. Concurrent other antitumor therapies;
4. Neoadjuvant therapy;
5. Subjects who have experienced a severe infection within one month before enrollment, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.;
6. Subjects with any active infection or unexplained fever > 38.5°C occurring during the screening period or before the first dose;
7. Presence of severe cardiovascular diseases: Grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval male ≥ 450 ms, female ≥ 470 ms); NYHA Class III-IV heart failure (according to the New York Heart Association classification, see Appendix 3), or echocardiogram indicating left ventricular ejection fraction (LVEF) < 50%;
8. History of other malignancies within the past five years (except for completely treated in situ cervical cancer or basal cell carcinoma or squamous cell carcinoma of the skin);
9. History of substance abuse involving psychiatric drugs that cannot be discontinued or presence of mental disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months
  Progression-Free Survival, is defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first after 6 months of treatment.

SECONDARY OUTCOMES:
LRC | 18 months
  Local Regional Control, is defined as the time from random assignment to documented local or regional relapse, whichever occurred first.
OS | 18 months
  Overall Survival, is defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
DMFS | 18 months
  Distant-Metastasis Free Survival, is defined as the time from random assignment to distant metastasis, or death from any cause, whichever occurred first.
PFS | 18 months
  Progression-Free Survival, is defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

OTHER OUTCOMES:
safety and toxicity | 18 months
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Y Zhang, Study Chair — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
only if researchers asked by email